CLINICAL TRIAL: NCT04353037
Title: PATCH 2 & 3: (Prevention and Treatment of COVID-19 With Hydroxychloroquine) A Double-blind Placebo Controlled Randomized Trial of Hydroxychloroquine in the Prevention and Treatment of COVID-19
Brief Title: PATCH 2&3:Prevention & Treatment of COVID-19 (Severe Acute Respiratory Syndrome Coronavirus 2) With Hydroxychloroquine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: As enrollment began external studies called into question the safety and efficacy of hydroxychloroquine as a treatment which resulted in controversy. The timing of the controversy significantly impacted our ability to enroll and retain participants.
Sponsor: UnitedHealth Group (Industry)
Collaborators: ProHealth Care Associates (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Dr. Deneen Vojta, Chief Medical Officer, Research and Development, UnitedHealth Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-0003
Record Dates: First submitted 2020-04-09; First posted 2020-04-20 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Coronavirus; Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Treatment and prevention study
Who Masked: Participant, Care Provider
Masking Description: For PATCH 2: participant and care provider are blinded. For PATCH 3: Health care worker is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sub Study 1 Patients (Experimental): Patients tested for COVID-19 who meet symptomology and age requirements for eligibility
  Interventions: Drug: Group 1 HCQ; Drug: Group 2 Placebo
- Sub Study 2 Health Care Workers (Experimental): Rate of COVID-19 infection (confirmed by accepted testing methods) at 2 months
  Interventions: Drug: Group 1 HCQ; Drug: Group 2 Placebo

INTERVENTIONS:
Drug: Group 1 HCQ — Enrolled participants randomized in Group 1 receive the HCQ drug
  Other Names: HCQ Group
Drug: Group 2 Placebo — Enrolled participants randomized in Group 2 will receive a placebo drug
  Other Names: Placebo Group

SUMMARY:
The proposed hypothesis is that high doses of hydroxychloroquine (HCQ) for at least 2 weeks can be effective antiviral medication both as a treatment in ambulatory patients and prophylaxis/treatment in health care workers because it impairs lysosomal function and reorganizes lipid raft (cholesterol and sphingolipid rich microdomains in the plasma membrane) content in cells, which are both critical determinants of Emerging Viral Disease (EVD) infection. This hypothesis is based on a growing literature linking chloroquine to antiviral activity. It is estimated that enough information exists to launch a clinical trial of hydroxychloroquine for COVID-19.

DETAILED DESCRIPTION:
Sub-Study 1: COVID-19 patients in self-quarantine. Group 1: Hydroxychloroquine 400 mg bid (two 200 mg tablets taken twice a day; totaling 800 mg per day) for two weeks; Group 2: Placebo 2 pills twice a day for two weeks

Sub-Study 2: Asymptomatic health care worker prophylaxis. Group 1: Hydroxychloroquine 600 mg once a day (three 200 mg tablets taken once a day) for up to 2 months; Group 2: Placebo 3 pills once a day for up to 2 months; cross-over from placebo to HCQ 600 mg once a day is allowed upon confirmatory diagnosis for COVID-19.

PRIMARY OBJECTIVES:

Sub-Study 1 (Patients tested for COVID-19 who meet symptomology and age requirements for eligibility): Rate of hospitalization

Sub-Study 2 (Health Care Workers): Rate of COVID-19 infection (confirmed by accepted testing methods) at 2 months

SECONDARY OBJECTIVES Sub-Study 1: Rate of secondary infection of co-inhabitants, adverse events, and negative for COVID-19 (confirmed by accepted testing methods) at 14 days

Sub-Study 2: Number of shifts missed; rate of adverse events, and hospitalization at 2 months

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Subjects meeting the following criteria by Sub-Study:

Sub-Study 1: 50-75 years of age; self-reporting as having a fever within four days prior to time of enrollment; and not requiring hospitalization. Enrolled individuals will undergo testing for COVID-19 and sent home for self-quarantine.Participant must be willing and able to provide informed consent, agree to testing for COVID-19 at time of enrollment to confirm diagnosis and two weeks at the end of treatment.

Sub-Study 2: Currently employed as a health care worker. Health care workers are defined as :

* Medical Doctor (MD)
* Doctor of Osteopathic Medicine (DO)
* Nurse Practitioner (NP)
* Physician's Assistant (PA)
* Registered Nurse (RN)
* other members of the medical care team with significant COVID-19 exposure;

Health care workers meeting the following criteria:

* asymptomatic and presumed negative for COVID-19 (no confirmatory testing conducted);
* scheduled for an average of >20 hours per week of clinical care over the next 2 months.

Participant must agree to standard clinical guidelines and undergo COVID-19 testing upon the presentation of symptoms indicative of an influenza like illness; if a confirmatory COVID-19 diagnosis is given, participant will be offered to cross-over to HCQ 600 mg qd.

* Willing to report compliance with HCQ in the form of a diary and participate in other forms of self-reporting (e.g., symptom tracker and experience log).
* Subjects are willing and able to go to designated areas for testing of COVID-19/SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2).
* Participants must be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Participants must have adequate baseline organ function

Exclusion Criteria:

* Inclusion Criteria

  * Able to give informed consent
  * Subjects meeting the following criteria by Sub-Study:

Sub-Study 1: 50-75 years of age; self-reporting as having a fever within four days prior to time of enrollment; and not requiring hospitalization. Enrolled individuals will undergo testing for COVID-19 and sent home for self-quarantine. Participant must be willing and able to provide informed consent, agree to testing for COVID-19 at time of enrollment to confirm diagnosis and two weeks at the end of treatment.

Sub-Study 2: Currently employed as a health care worker (Medical Doctor, MD; Doctor of Osteopathic Medicine, DO; Nurse Practitioner, NP; Physician's Assistant, PA; and Registered Nurse, RN or other members of the medical care team with significant COVID-19 exposure); asymptomatic and presumed negative for COVID-19 (no confirmatory testing conducted); scheduled for an average of >20 hours per week of clinical care over the next 2 months. Participant must agree to standard clinical guidelines and undergo COVID-19 testing upon the presentation of symptoms indicative of an influenza like illness; if a confirmatory COVID-19 diagnosis is given, participant will be offered to cross-over to HCQ 600 mg qd.

* Willing to report compliance with HCQ in the form of a diary and participate in other forms of self-reporting (e.g., symptom tracker and experience log).
* Subjects are willing and able to go to designated areas for testing of COVID-19/SARS-CoV-2.
* Participant must be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Participant must have adequate baseline organ function

Exclusion Criteria

* Allergy to hydroxychloroquine
* Pregnant or lactating or positive pregnancy test during pre-medication examination
* Receiving any trial treatment drug for 2019-ncov within 14 days prior to screening evaluation (off label, compassionate use or trial related).
* Known retinal disease including but not limited to macular degeneration, retinal vein occlusion, visual field defect, diabetic retinopathy
* History of interstitial lung disease or chronic pneumonitis unrelated COVID-19.
* Due to risk of disease exacerbation, participants with porphyria or psoriasis are ineligible unless the disease is well-controlled, and they are under the care of a specialist for the disorder who agrees to monitor the Participant for exacerbations.
* Participants with serious intercurrent illness that requires active intravenous therapy, intense monitoring, or frequent dose adjustments for medication including but not limited to infectious disease, cancer, autoimmune disease, cardiovascular disease.
* Participants who have undergone major abdominal, thoracic, spine or central nervous system (CNS) surgery in the last 2 months, or plan to undergo surgery during study participation.
* Participants receiving cytochrome P450 enzyme-inducing anticonvulsant drugs (i.e. phenytoin, carbamazepine, Phenobarbital, primidone or oxcarbazepine) within 4 weeks of the start of the study treatment
* Participants currently taking digoxin
* History or evidence of increased cardiovascular risk including any of the following:
* Left ventricular ejection fraction (LVEF) < institutional lower limit of normal. Baseline echocardiogram is not required.
* Current clinically significant uncontrolled arrhythmias. Exception: Subjects with controlled atrial fibrillation
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to enrollment
* Current ≥ Class II congestive heart failure as defined by New York Heart Association.
* Deemed unable to participate for medical reasons identified by Co-PI and study staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deneen Vojta, MD, Principal Investigator — UnitedHealth Group
Locations (1):
- ProHealth New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected and managed by Optumcare and UnitedHealth Group Research & Development. Redacted/aggregate data will be shared with the University Of Penn using approved data sharing protocols.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year

REFERENCES:
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Ong SWX, Tan YK, Chia PY, Lee TH, Ng OT, Wong MSY, Marimuthu K. Air, Surface Environmental, and Personal Protective Equipment Contamination by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) From a Symptomatic Patient. JAMA. 2020 Apr 28;323(16):1610-1612. doi: 10.1001/jama.2020.3227. PMID 32129805
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Liu J, Liao X, Qian S, Yuan J, Wang F, Liu Y, Wang Z, Wang FS, Liu L, Zhang Z. Community Transmission of Severe Acute Respiratory Syndrome Coronavirus 2, Shenzhen, China, 2020. Emerg Infect Dis. 2020 Jun;26(6):1320-1323. doi: 10.3201/eid2606.200239. Epub 2020 Jun 17. PMID 32125269
- [Background] Li F. Receptor recognition mechanisms of coronaviruses: a decade of structural studies. J Virol. 2015 Feb;89(4):1954-64. doi: 10.1128/JVI.02615-14. Epub 2014 Nov 26. PMID 25428871
- [Background] Wang H, Yang P, Liu K, Guo F, Zhang Y, Zhang G, Jiang C. SARS coronavirus entry into host cells through a novel clathrin- and caveolae-independent endocytic pathway. Cell Res. 2008 Feb;18(2):290-301. doi: 10.1038/cr.2008.15. PMID 18227861
- [Background] Chu VC, McElroy LJ, Chu V, Bauman BE, Whittaker GR. The avian coronavirus infectious bronchitis virus undergoes direct low-pH-dependent fusion activation during entry into host cells. J Virol. 2006 Apr;80(7):3180-8. doi: 10.1128/JVI.80.7.3180-3188.2006. PMID 16537586
- [Background] Zheng Y, Shang J, Yang Y, Liu C, Wan Y, Geng Q, Wang M, Baric R, Li F. Lysosomal Proteases Are a Determinant of Coronavirus Tropism. J Virol. 2018 Nov 27;92(24):e01504-18. doi: 10.1128/JVI.01504-18. Print 2018 Dec 15. PMID 30258004
- [Background] Keyaerts E, Li S, Vijgen L, Rysman E, Verbeeck J, Van Ranst M, Maes P. Antiviral activity of chloroquine against human coronavirus OC43 infection in newborn mice. Antimicrob Agents Chemother. 2009 Aug;53(8):3416-21. doi: 10.1128/AAC.01509-08. Epub 2009 Jun 8. PMID 19506054
- [Background] Vincent MJ, Bergeron E, Benjannet S, Erickson BR, Rollin PE, Ksiazek TG, Seidah NG, Nichol ST. Chloroquine is a potent inhibitor of SARS coronavirus infection and spread. Virol J. 2005 Aug 22;2:69. doi: 10.1186/1743-422X-2-69. PMID 16115318
- [Background] de Wilde AH, Jochmans D, Posthuma CC, Zevenhoven-Dobbe JC, van Nieuwkoop S, Bestebroer TM, van den Hoogen BG, Neyts J, Snijder EJ. Screening of an FDA-approved compound library identifies four small-molecule inhibitors of Middle East respiratory syndrome coronavirus replication in cell culture. Antimicrob Agents Chemother. 2014 Aug;58(8):4875-84. doi: 10.1128/AAC.03011-14. Epub 2014 May 19. PMID 24841269
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Amaravadi RK, Lippincott-Schwartz J, Yin XM, Weiss WA, Takebe N, Timmer W, DiPaola RS, Lotze MT, White E. Principles and current strategies for targeting autophagy for cancer treatment. Clin Cancer Res. 2011 Feb 15;17(4):654-66. doi: 10.1158/1078-0432.CCR-10-2634. PMID 21325294
- [Background] Rangwala R, Chang YC, Hu J, Algazy KM, Evans TL, Fecher LA, Schuchter LM, Torigian DA, Panosian JT, Troxel AB, Tan KS, Heitjan DF, DeMichele AM, Vaughn DJ, Redlinger M, Alavi A, Kaiser J, Pontiggia L, Davis LE, O'Dwyer PJ, Amaravadi RK. Combined MTOR and autophagy inhibition: phase I trial of hydroxychloroquine and temsirolimus in patients with advanced solid tumors and melanoma. Autophagy. 2014 Aug;10(8):1391-402. doi: 10.4161/auto.29119. Epub 2014 May 20. PMID 24991838
- [Background] Rangwala R, Leone R, Chang YC, Fecher LA, Schuchter LM, Kramer A, Tan KS, Heitjan DF, Rodgers G, Gallagher M, Piao S, Troxel AB, Evans TL, DeMichele AM, Nathanson KL, O'Dwyer PJ, Kaiser J, Pontiggia L, Davis LE, Amaravadi RK. Phase I trial of hydroxychloroquine with dose-intense temozolomide in patients with advanced solid tumors and melanoma. Autophagy. 2014 Aug;10(8):1369-79. doi: 10.4161/auto.29118. Epub 2014 May 20. PMID 24991839
- [Background] Vogl DT, Stadtmauer EA, Tan KS, Heitjan DF, Davis LE, Pontiggia L, Rangwala R, Piao S, Chang YC, Scott EC, Paul TM, Nichols CW, Porter DL, Kaplan J, Mallon G, Bradner JE, Amaravadi RK. Combined autophagy and proteasome inhibition: a phase 1 trial of hydroxychloroquine and bortezomib in patients with relapsed/refractory myeloma. Autophagy. 2014 Aug;10(8):1380-90. doi: 10.4161/auto.29264. Epub 2014 May 20. PMID 24991834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sub study 1 HCQ & Placebo groups were identified as patient at least 50 years old self-reported as having a fever within the last four days will undergo swab testing for COVID-19, and then sent home for a self-imposed quarantine that will end 14 days from the start of treatment and consenting patients were randomized. Sub study 2 HCQ and Placebo groups were recruited first through completion of an interest questionnaire then contacted by study PI or designee to assess eligibility consent.
Pre-assignment Details: If Sub Study 1 patients received a negative PCR-test then they were considered no longer a part of the study and had a conversation with the PI or designee. Recruitment was done this way because early in the pandemic, time to receive PCR test results was unclear. At study conclusion 9 substudy 1 participants were Covid positive. 6 of those Covid positive participants completed the study. 30 participants from sub study 2 met eligibility criteria with 13 participants completing the full study.
Groups:
- Sub Study 1 Group 1 (HCQ): COVID-19 positive PCR patients in self-quarantine randomized to this arm will be treated with hydroxychloroquine 400mg twice a day for 14 days.
- Sub Study 1 Group 2 (Placebo): COVID-19 positive PCR patients in self-quarantine randomized to this arm will be treated with placebo 2 pills twice a day for 14 days.
- Sub Study 2 Group 1 (HCQ): Currently employed as a health care worker. Must be asymptomatic and presumed negative for COVID-19. Health care workers randomized into this arm will be treated with hydroxychloroquine 600 mg qd (three 200 mg tablets taken once a day) for 2 months.
- Sub Study 2 Group 2 (Placebo): Currently employed as a health care worker. Must be asymptomatic and presumed negative for COVID-19. Health care workers randomized into this arm will be treated with Placebo pills (three 200 mg tablets taken once a day) for 2 months.
Period: Overall Study
Arm/Group | Sub Study 1 Group 1 (HCQ) | Sub Study 1 Group 2 (Placebo) | Sub Study 2 Group 1 (HCQ) | Sub Study 2 Group 2 (Placebo)
Started | 6 | 3 | 13 | 17
Completed | 6 | 0 | 6 | 7
Not Completed | 0 | 3 | 7 | 10
Not completed — Lost to Follow-up | 0 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 5
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Exposure Change | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All eligible randomized patients
Groups:
- Substudy 1 Group 1 (HCQ): COVID-19 positive PCR patients aged 50-75 in self-quarantine randomized to this arm will be treated with hydroxychloroquine 400mg twice a day for 14 days.
- Substudy 1 Group 2 (Placebo): COVID-19 positive PCR patients aged 50-75 in self-quarantine randomized to this arm will be treated with placebo 2 pills twice a day for 14 days.
- Substudy 2 Group 1 (HCQ): Currently employed as a health care worker aged 18 or older. Must be asymptomatic and presumed negative for COVID-19.
  Health care workers randomized into this arm will be treated with hydroxychloroquine 600 mg daily (three 200 mg tablets taken once a day) for 2 months.
- Substudy 2 Group 2 (Placebo): Currently employed as a health care worker aged 18 or older. Must be asymptomatic and presumed negative for COVID-19.
  Health care workers randomized into this arm will be treated with Placebo pills (three 200 mg tablets taken once a day) for 2 months.
- Total: Total of all reporting groups
Arm/Group | Substudy 1 Group 1 (HCQ) | Substudy 1 Group 2 (Placebo) | Substudy 2 Group 1 (HCQ) | Substudy 2 Group 2 (Placebo) | Total
Number analyzed (Participants) | 6 | 3 | 13 | 17 | 39
Age, Continuous [Median (Full Range); unit: years] | 59 [54 to 68] | 58 [56 to 61] | 45 [34 to 61] | 49 [31 to 66] | 49 [31 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 8 | 11 | 23
  Male | 3 | 2 | 5 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 5 | 1 | 13 | 17 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 2
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 4 | 0 | 10 | 11 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Substudy 1 - Number of COVID-19+ PCR Patients in Self-quarantine Who Are Hospitalized
Description: Number of COVID-19+ PCR patients in self-quarantine who are hospitalized up to 31 days after beginning HCQ or Placebo
Time Frame: Until completion of study, 29 to 31 days after beginning treatment.
Population: Evaluable for primary outcome, having completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub Study 1 Group 1 (HCQ) | Sub Study 1 Group 2 (Placebo)
Number analyzed (Participants) | 6 | 0
Participants | 0 | 0

2. Primary Outcome: Sub Study 2:Number of Health Care Workers Testing Positive at 2 Months
Description: Rate of COVID-19 infection (confirmed by accepted testing methods) at 2 months
Time Frame: Until completion of study, 2 months after start of treatment.
Population: Evaluable for primary outcome, having completed the study.
Measure: Count of Participants; unit: Participants
Groups:
- Sub Study 2 Group 1 (HCQ): Currently employed as a health care worker. Must be asymptomatic and presumed negative for COVID-19. Health care workers randomized into this arm will be treated with hydroxychloroquine 600 mg daily (three 200 mg tablets taken once a day) for 2 months.
Arm/Group | Sub Study 2 Group 1 (HCQ) | Sub Study 2 Group 2 (Placebo)
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

3. Secondary Outcome: Sub Study 1 - Secondary Infection of Co-inhabitants of COVID-19 Positive PCR Patients in Self-quarantine
Description: Co-inhabitants of COVID-19 positive PCR patients in self-quarantine that test positive up to 31 days after patient begins treatment with HCQ or Placebo
Time Frame: Until completion of study, 29 to 31 days after beginning treatment.
Population: Co-inhabitants of patients evaluable for primary outcome, who completed the study. There were 16 co-inhabitants of the Sub study 1 Group 1 (HCQ).
Measure: Count of Participants; unit: Participants
Arm/Group | Sub Study 1 Group 1 (HCQ) | Sub Study 1 Group 2 (Placebo)
Number analyzed (Participants) | 16 | 0
Participants | 0 | 0

4. Secondary Outcome: Sub Study 1 - Rate of Negative Tests at End of Treatment for COVID-19 Positive PCR Patients in Self-quarantine
Description: Rate of negative tests at end of treatment for COVID-19 positive PCR patients in self-quarantine
Time Frame: 15-17 days after completion of 14 day treatment
Population: Evaluable for primary outcome, having completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub Study 1 Group 1 (HCQ) | Sub Study 1 Group 2 (Placebo)
Number analyzed (Participants) | 6 | 0
Participants | 6 | 0

5. Secondary Outcome: Sub Study 1 - Rate of Negative Tests at End of Treatment for COVID-19 Positive PCR Patients in Self-quarantine
Description: Rate of negative tests at end of treatment for COVID-19 positive PCR patients in self-quarantine
Time Frame: 1-3 days after completion of 14 day treatment
Population: Evaluable for primary outcome, having completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub Study 1 Group 1 (HCQ) | Sub Study 1 Group 2 (Placebo)
Number analyzed (Participants) | 6 | 0
Participants | 4 | 0

6. Secondary Outcome: Sub Study 2:Health Care Workers:Number of Shifts Missed
Description: Any work time missed because the participant experienced COVID-like symptoms during their active 2 month period
Time Frame: up to ~60 days after enrollment
Population: We had no positive Covid-19 tests for Sub Study 2 healthcare workers so we couldn't measure this outcome.
Arm/Group | Sub Study 2 Group 1 (HCQ) | Sub Study 2 Group 2 (Placebo)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Sub Study 2:Health Care Workers: Assessment of Any Medical Events That Occur During the ~60 Day Active Period
Description: Assessment of any medical events that occur during the ~60 day active period that is felt to be related to receipt of HCQ
Time Frame: Until completion of study, 2 months (~60 days) after start of treatment.
Population: Evaluable for primary outcome, having completed the study or removed from study due to moderate or more serious adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | Sub Study 2 Group 1 (HCQ) | Sub Study 2 Group 2 (Placebo)
Number analyzed (Participants) | 8 | 7
Participants
  moderate adverse events | 2 | 0
  minor adverse events | 1 | 0

8. Secondary Outcome: Sub Study 2:Health Care Workers:Rate of Hospitalization
Description: if the participant gets COVID and has severe symptoms and hospitalized, end point reached if before the end of the 2 month period
Time Frame: Until completion of study, 2 months after start of treatment.
Population: Evaluable for primary outcome, having completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub Study 2 Group 1 (HCQ) | Sub Study 2 Group 2 (Placebo)
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Until completion of study, 2 months after start of treatment.
Description: No adverse events were reported for Sub study 1. For SubStudy 2 group 1, 6 participants completed and were evaluable for primary outcomes, 2 participants were removed from study due to moderate or serious adverse event prior to meeting the evaluable benchmark.
Groups:
- Sub Study 1 Group 1 (HCQ): COVID-19+ PCR patients in self-quarantine randomized to this arm will be treated with hydroxychloroquine 400mg bid for 14 days.
- Sub Study 1 Group 2 (Placebo): COVID-19+ PCR patients in self-quarantine randomized to this arm will be treated with Place 2 pills bid for 14 days.
Arm/Group | Sub Study 1 Group 1 (HCQ) | Sub Study 1 Group 2 (Placebo) | Sub Study 2 Group 1 (HCQ) | Sub Study 2 Group 2 (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 3/8 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub Study 1 Group 1 (HCQ) (N=6) | Sub Study 1 Group 2 (Placebo) (N=3) | Sub Study 2 Group 1 (HCQ) (N=8) | Sub Study 2 Group 2 (Placebo) (N=7)
Nasal congestion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild Nasal congestion
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Moderate Headache over a period of 6 days
Angioedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Moderate Swelling of face (angioedema) over a period of 1 day.
Nausea (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Moderate Nausea over a period of 6 days
Decreased Appetite (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — moderate decreased appetite over a period of 6 days
abdominal pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — moderate abdominal pain over a period of 6 days

LIMITATIONS AND CAVEATS:
No healthcare workers had a positive Covid test during the study period so the outcome for missed shifts due a positive Covid result was not measured.

Due to low enrollment numbers, only a descriptive analysis was reported and we did not test any of the hypotheses described in the statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04353037/Prot_SAP_000.pdf